CLINICAL TRIAL: NCT00005056
Title: A Phase II Trial of Bryostatin-1 in Hypernephroma
Brief Title: Bryostatin 1 In Treating Patients With Progressive Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CRC-PHASE-I/II-PH2/034; CDR0000067651 (Registry Identifier: PDQ (Physician Data Query)); EU-20001; NCI-T95-0024
Record Dates: First submitted 2000-04-06; First posted 2004-08-09 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2006-06

CONDITIONS: Kidney Cancer
Keywords: stage I renal cell cancer; stage II renal cell cancer; stage III renal cell cancer; stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — bryostatin 1

INTERVENTIONS:
Drug: bryostatin 1

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of bryostatin 1 in treating patients who have progressive kidney cancer

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rates in patients with progressive hypernephroma treated with bryostatin 1. II. Determine the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study. Patients receive bryostatin 1 IV over 24 hours on days 1, 8, and 15. Treatment repeats every 4 weeks for 2 courses. For patients with stable or responding disease after completion of course 2, treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 14-25 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven progressive hypernephroma Bidimensionally measurable disease with documented progression within 2 months prior to study entry Sites of measurable or evaluable disease must be outside prior radiation ports No active symptomatic CNS disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: WHO 0-2 Life expectancy: Greater than 3 months Hematopoietic: Granulocyte count greater than 1,500/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin less than 1.17 mg/dL SGOT or SGPT less than 2.5 times normal Renal: Creatinine less than 1.70 mg/dL Other: No other prior or concurrent malignancy except adequately treated cone biopsied carcinoma in situ of the cervix or basal cell or squamous cell skin cancer No severe or uncontrolled nonmalignant systemic disease that would make the patient a poor medical risk No uncontrolled active infection Not pregnant or nursing Fertile patients must use effective contraception during and for 4 weeks after study

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior immunotherapy and recovered Chemotherapy: No prior chemotherapy Endocrine therapy: At least 4 weeks since prior endocrine therapy or steroids and recovered No concurrent systemic steroids Radiotherapy: See Disease Characteristics At least 4 weeks since prior radiotherapy and recovered No concurrent radiotherapy Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-03; Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian L. Harris, MD, Study Chair — Oxford University Hospitals NHS Trust
Locations (2):
- United Kingdom (2):
  - Oxford Radcliffe Hospital, Oxford, England
  - Imperial Cancer Research Fund Medical Oncology Unit, Oxford, England